CLINICAL TRIAL: NCT06887764
Title: A Pilot Study to Examine the Effect of a Powered Knee Orthosis on Crouch Gait in Cerebral Palsy
Brief Title: Robotic Knee Orthosis-assisted Walking in CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Principal Investigator, David Scher, MD, Attending Orthopaedic Surgeon, Hospital for Special Surgery, New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-2299
Record Dates: First submitted 2025-03-07; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Crouch Gait; Cerebral Palsy (CP)
Keywords: Robotic Knee Orthosis; Crouch Gait; Flexed-knee Gait; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect of a powered knee orthosis in individuals with Cerebral Palsy and Flexed-knee Gait (Experimental)
  Interventions: Device: RKO-assisted walking in children with CP

INTERVENTIONS:
Device: RKO-assisted walking in children with CP — The investigators will assess walking in each of the following conditions: shod (shoes or shoes + AFO) and RKO-assisted (shoes + RKO), to achieve the following: (1) Evaluate the effect of RKO, compared to shod upon endurance in children with CP at GMFCS level II, and (2) Evaluate the effect of RKO, compared to shod, upon temporal-spatial parameters, lower limb sagittal joint kinematics, and muscle EMG in children with CP at GMFCS level II.

SUMMARY:
Robotic exoskeletons are becoming increasingly accepted to provide upright mobility in individuals with neurological disorders. These devices can assist in overcoming gravitational forces and reduce energy consumption. Agilik is one such device intended for children with neurological disorders. However, Agilik is relatively new, and its efficacy in children with CP is unknown. Therefore, this study aims to assess the effectiveness of Agilik as an assistive device for children with CP and crouch gait. In this pilot study, ten children with CP, GMFCS level II, and crouch gait will walk with Agilik under the supervision of a physical therapist. Assessments of walking with AFO and Agilik will evaluate the efficacy of the device. The pilot study will assess if Agilik decreases crouch and improves gait characteristics in children with CP.

DETAILED DESCRIPTION:
Robotic knee orthosis (RKO) can assist with voluntary knee extension and potentially reduce crouch/flexed-knee gait, but the efficacy of this technology in children with CP is unknown. This study aims to assess the effectiveness of Agilik as an assistive device for children with CP. Ten children with CP, ages 8 to 17 years, and at GMFCS level II, will be recruited for this pilot study. Each child will participate in a total of four visits over four weeks duration. The first three visits will also include RKO device fitting and tuning, followed by RKO-assisted walking practice to help with device acclamation. The walking practice will last up to 30 minutes. A two-minute walk test (2MWT) will be conducted at the first visit, which will serve as a reference to assess any shift in endurance from device-tuning/practice visits. The fourth and final visit will include 2MWT and 3D motion capture of shod and RKO-assisted conditions and may take up to 3 to 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cerebral palsy at GMFCS level II
* Exhibits crouch gait
* Between 8 to 17 years of age
* Hip flexion contracture less than 5 degrees
* Knee flexion contracture less than 20 degrees when measured in prone with hips extended
* Thigh-foot angle is between 10 degrees (internal) to 25 degrees (external) in prone
* Can walk a minimum distance of 10 meters without stopping

Exclusion Criteria:

* Plantarflexion contracture, when measured in neutral foot alignment
* No other neurological, musculoskeletal, or cardiorespiratory health conditions or injuries
* The presence of any cognitive impairment that could limit the ability to understand, follow simple directions, and inform when in pain
* Inability to participate in the study because of recent orthopedic surgery (within twelve months) or botox intervention (within six months)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Distance from 2MWT | From enrollment until data collection is performed, 4 weeks after enrollment
  The distance covered by participants during a two-minute walking test (2MWT) will be compared between RKO-assisted and shod conditions.
Step length | At the end of study visit for each participant, approximately 4 weeks from enrollment
  Mean step length (distance between the two feet measured from the heel of one foot to the heel of the contralateral foot while both feet are on the ground) during walking will be compared between RKO-assisted and shod conditions.
Single limb support time | At the end of study visit for each participant, approximately 4 weeks from enrollment
  Mean single limb support time (duration just one foot by itself is on the ground) during walking will be compared between RKO-assisted and shod conditions.
Walking speed | At the end of study visit for each participant, approximately 4 weeks from enrollment
  Mean walking speed during walking will be compared between RKO-assisted and shod conditions.
Lower limb joint kinematics | At the end of study visit for each participant, approximately 4 weeks from enrollment
  The sagittal plane lower limb joint angles (degrees) during walking will be compared to evaluate the difference between RKO-assisted and shod conditions.
Binary indicator of improvement in walking distance with RKO use | At the end of study visit for each participant, approximately 4 weeks from enrollment
  "Yes" if the walking distance in the RKO-assisted condition was greater than shod, and "No" if there was no improvement.
Lower limb electromyography data | At the end of study visit for each participant, approximately 4 weeks from enrollment
  Electromyography (EMG) amplitude and duration of lower limb anti-gravity muscles (rectus femoris, vastus lateralis, vastus medialis, medial gastrocnemius, soleus, and gluteus maximus) will be compared between RKO-assisted and shod conditions. The EMG data will be filtered and rectified to compute linear envelopes. From these envelopes, the average value of EMG amplitude and duration will be compared between RKO-assisted and shod conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The study results (de-identified) will be disseminated in conference abstracts and peer-reviewed journal articles.
Supporting Information: Study Protocol, SAP
Time Frame: Within 12 months of the trial completion.
Access Criteria: Data and supporting information will be shared upon reasonable request to the PI. After the PI reviews and approves the applicant's request, de-identified information will be provided.